CLINICAL TRIAL: NCT06237413
Title: A Phase I/II Dose Escalation Study to Evaluating the Tolerability, Safety, Efficacy and Pharmacokinetics of ZG2001 Tosilate Tablets in Participants With KRAS Mutated Advanced Solid Tumours
Brief Title: A Study of ZG2001 in Participants With KRAS Mutated Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG2001-001
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Solid Tumor; KRAS Mutation-Related Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Dose Escalation (Experimental): This Phase adopts an open-label design, with an Accelerated Titration(AT) design for the low-dose group (50 mg Bid) and the standard "3+3" design for the high-dose groups（100 mg Bid、50 mg Qd、100 mg Qd、200 mg Qd）.
  Interventions: Drug: ZG2001 Tosilate Tablets
- Phase 2 Dose Expansion (Experimental): After the completion of the dose escalation study, RP2D will be selected for dose expansion in advanced solid tumors (such as non-small cell lung cancer, colorectal cancer, pancreatic cancer, etc.) with KRAS mutations that have failed at least the first-line standard treatment
  Interventions: Drug: ZG2001 Tosilate Tablets

INTERVENTIONS:
Drug: ZG2001 Tosilate Tablets — ZG2001 will be administered orally once or twice daily in a continuous regimen
  Other Names: ZG2001

SUMMARY:
This study will evaluate the tolerability, safety, effects, and pharmacokinetics of ZG2001 in Participants with advanced solid tumors that have a KRAS mutation.

ELIGIBILITY:
Inclusion Criteria:

* Participants who fully understood this study and voluntarily signed the informed consent form;
* Men or women ≥ 18 years old;
* Participants with a KRAS mutant solid tumor should have progressed on or are ineligible for all therapy(ies) known to confer clinical benefit.
* ECOG Performance Status (PS) 0 or 1;
* Life expectancy > 3 months.

Exclusion Criteria:

* Received any SOS1 inhibitors;
* Participants with a known history of hypersensitivity reactions to the ingredients of the preparations used in this study;
* Other conditions that the investigator considers to be unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-08-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 21 Days
  A DLT is defined as any Grade ≥ 3 AE meeting the criteria listed below occurring during the 1st treatment cycle of ZG2001 (Day 1 through Day 21) where the relationship to ZG2001 cannot be ruled out.
Incidence of Treatment-Emergent Adverse Events | Up to 24 Months
  Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No